CLINICAL TRIAL: NCT01990222
Title: Leveraging Mobile Health Technology to Optimize Early Stimulant Medication Treatment: A Feasibility Pilot
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Bonnie Zima, MD MPH, Associate Director of the Jane and Terry Semel Institute's Health Services Research Center and Professor-in-Residence in the UCLA Department of Psychiatry and Behavioral Sciences at the David Geffen School of Medicine, University of California, Los Angeles
Other Study IDs: UL1TR000124 (NIH); IRB#12-001879 (Other: University of California at Los Angeles (UCLA) IRB)
Record Dates: First submitted 2013-07-01; First posted 2013-11-21 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of this study is to develop and test a mobile web application to optimize early stimulant medication treatment for children receiving care for Attention/Deficit Hyperactivity Disorder (ADHD) in a publicly-funded mental health clinic.

DETAILED DESCRIPTION:
In other words, the study will find out whether it is feasible and acceptable for parents to receive reminders for clinic visits and ADHD medication and enter daily ratings of their child's ADHD symptoms and medication side effects into a smart phone. It will also examine whether it is feasible and acceptable for doctors to use this information summarized on a tablet (iPad) screen during a medication follow-up visit. If the parent consents, the study will also examine whether it is feasible and acceptable for the child's teacher to enter their ratings of ADHD symptoms twice a week using a link on their email. This information will also be included in the doctor's iPad screen. If this technology is found to be promising, then a larger study will be done to examine if medication treatment is safer, more consistent, and more effective using this technology compared to usual care. This is important because the technology may remove the burden on parents and teachers to report ADHD symptoms and medication side effects using paper forms, and for doctors to record this information in the medical record. In total, there will be 12 parent/ child dyads, 6 clinicians and up to 12 teachers enrolled. Each parent/child dyad will be videotaped for up to 3 visits with the clinician (n=36 videotaped sessions). The study time period is from the first visit that ADHD medication is prescribed to the time of the third follow-up medication visit. We anticipate that the follow-up visits will be every 1-2 weeks during this early phase of stimulant medication treatment. Thus, the study time period for each parent/child dyad will be between 4-8 weeks. We anticipate that data collection will occur between August 19, 2013 and June 31, 2014.

ELIGIBILITY:
Inclusion Criteria:

* parent's and child's primary language is English or Spanish
* child is between 5-11 years
* child received a clinical diagnosis of ADHD
* child is receiving stimulant medication for the first time
* child does not take any other medication on a regular basis (like every day)

Exclusion Criteria:

* any chronic medical condition that requires on-going medication management
* prescription of combined psychotropic medication
* moderate-severe developmental delays, mental retardation or autism

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Parents taking their children to Augustus Hawkins Mental Health Center for treatment of ADHD who were prescribed stimulant medication for the first time. The attending physicians will work at the clinic.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Stimulant medication adherence | medication follow-up visit 1- visit 3, approx 8 weeks, depending on scheduling of the 3 med visits, usually 1 every 2 weeks
  parent-reported stimulant medication adherence

SECONDARY OUTCOMES:
Parent-provider communication | Once every two weeks for each participant, over approx 8 weeks, depending on scheduling of the 3 med visits, usually 1 every 2 weeks
  Each parent/child dyad, if consented, will have their first three medication visits with their doctor videotaped. These visits are typically once every two weeks for each dyad.
Clinic follow-up visit attendance | medication follow-up visit 1-visit 3, approx 8 weeks, depending on scheduling of the 3 med visits, usually 1 every 2 weeks
  attendance of scheduled follow-up clinic visits for medication management

OTHER OUTCOMES:
Parent-centered medication management | between medication follow-up visit 1- visit 3, over approx 8 weeks, depending on scheduling of the 3 med visits, usually 1 every 2 weeks
  stimulant medication treatment decisions that are responsive to parent- reported symptoms and medication side effects and treatment acceptability ratings

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie Zima, MD, MPH, Principal Investigator — University of California, Los Angeles
Locations (3):
- United States (3):
  - Augustus Hawkins Mental Health Center, Los Angeles, California
  - UCLA Children's Health Center, Los Angeles, California
  - Child and Family Guidance Center, Northridge, California